CLINICAL TRIAL: NCT07148375
Title: Anterograde Headless Screw Fixation For Treatment Of Medial Malleolar Fractures .
Brief Title: Fixation of Medial Malleolar Fractures .
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Abdelhakam, Anterograde headless screw fixation for treatment of medial malleolar fractures, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-8-1MS
Record Dates: First submitted 2025-08-21; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Anterograde Screw Fixation for Medial Malleolus Fractures

STUDY DESIGN:
Intervention Model Description: The aim of this study is to evaluate the functional and radiological outcomes following of fixation of Herscovici type B and type C medial malleolar fractures with anterograde headless screws.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Any patient with medial Malleolus fracture (Experimental): Anterograde herbert screws for fixation of medial Malleolus fractures
  Interventions: Procedure: Anterograde screws for medial Malleolus fractures

INTERVENTIONS:
Procedure: Anterograde screws for medial Malleolus fractures — Fixation of medial Malleolus fracures by anterograde headless screws

SUMMARY:
The aim of this study is to evaluate the functional and radiological outcomes following of fixation of Herscovici type B and type C medial malleolar fractures with anterograde headless screws.

DETAILED DESCRIPTION:
Ankle fracture is one of the most common orthopaedic injuries[1]. Medial Malleolus fractures are Classified According to Herscovici classification Using the anteroposterior (AP) radiograph, he described type A fractures as avulsions of the tip of the malleolus, type B occurring between the tip and the level of the tibial plafond, type C at the level of the plafond, and type D extending vertically above the plafond [2].

The aim of operative treatment in ankle fractures is to provide stable internal fixation and allow early movement . Several fixation techniques had been described for the anatomic reduction of fractures, including Kirschner wires (K-wire), tension band method, fixation with suture anchors, bioabsorbable screw fixation, a FiberWire loop with a tension band, and screw fixation[3].

In addition to these techniques, fixation with anterograde screws can also be used for medial malleolar fixation. Given that with time the size of the fractured distal fragment in a medial malleolar fracture is insufficient for retrograde fixation as ln Herscovici type B and type C[4].

Screws are commonly used to fix medial malleolus fractures , offering advantages like good compression and stability[5]. the advantage of the anterograde headless screw fixation technique over the other techniques is that less dissection of the deltoid ligament is required during fixation , no need for screws removal , less soft tissue irritation and less discomfort [6].

ELIGIBILITY:
Inclusion Criteria Patients with Isolted medial malleolar fractures or combined with other fractures [ bimalleolar or trimalleolar Fractures]

Individuals meeting the following criteria will be included in the study:

1. Patient Age between 20 _50 Years old.
2. Simple or compound fractures (Grade I).
3. Recent Fractures .
4. Herscovici Type B and C Fractures. a:

   -

   Exclusion Criteria:
   * Skeletally Immature . Compound fractures ( Grade II,III). Pathological fractures. Diabetic patients .

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Anterograde Headless Screw Fixation for Treatment of Medial Malleolar Fractures . | 1 year
  Ankle fracture is one of the most common orthopaedic injuries[1]. Medial Malleolus fractures are Classified According to Herscovici classification Using the anteroposterior (AP) radiograph, he described type A fractures as avulsions of the tip of the malleolus, type B occurring between the tip and the level of the tibial plafond, type C at the level of the plafond, and type D extending vertically above the plafond [2].
  The aim of operative treatment in ankle fractures is to provide stable internal fixation and allow early movement . Several fixation techniques had been described for the anatomic reduction of fractures, including Kirschner wires (K-wire), tension band method, fixation with suture anchors, bioabsorbable screw fixation, a FiberWire loop with a tension band, and screw fixation[3].
  In addition to these techniques, fixation with anterograde screws can also be used for medial malleolar fixation. Given that with time the size of the fractured distal fragment in a media

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided